CLINICAL TRIAL: NCT03325985
Title: Emergency Medicine Palliative Care Access (EMPallA)
Brief Title: Emergency Medicine Palliative Care Access
Acronym: EMPallA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Beaumont Health (Other); Dana-Farber/Brigham and Women's Cancer Center (Other); Ohio State University (Other); University of Florida (Other); Yale University (Other); Patient-Centered Outcomes Research Institute (Other); Hackensack Meridian Health (Other); Atlantic Health System (Other); University of California, Irvine (Other); University of California, San Diego (Other); University of California, Los Angeles (Other); Northwestern University (Other); Rush University (Other); Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-01211; R-1609-36306 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced Cancer; End Stage Organ Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led telephonic case management (Experimental): * Telephonic nurses will contact patients within 72 hours of enrollment
  * Patients will speak with the telephonic nurse over the phone once a week (or as often as needed) for a duration of 6 months.
  Interventions: Behavioral: Nurse-led telephonic case management
- Facilitated, outpatient specialty palliative care (Active Comparator): * Patients will be scheduled for their first in-person palliative care visit within two weeks of enrollment and then once a month for 6 months.
  * Clinic visits will be scheduled the same day as other specialty appointments if possible
  Interventions: Behavioral: Facilitated,outpatient specialty palliative care

INTERVENTIONS:
Behavioral: Nurse-led telephonic case management — Telephonic meetings with a palliative care nurse. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
  Arms: Nurse-led telephonic case management
Behavioral: Facilitated,outpatient specialty palliative care — In-person or telehealth palliative care visits with a palliative care provider. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
  Arms: Facilitated, outpatient specialty palliative care

SUMMARY:
This is a two-arm, multi-site randomized controlled trial of 1,350 older adults (50+ years) with either advanced cancer (defined as metastatic solid tumor) or poor prognosis end-stage organ failure (New York Heart Association (NYHA) Class III or IV Congestive Heart Failure (CHF), End-Stage Renal Disease (ESRD), defined as Glomerular Filtration Rate (GFR) < 15 ml/min/m2 or dialysis ; or Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage III or higher, or oxygen-dependent chronic obstructive pulmonary disease (COPD) who present to the Emergency Department (ED), along with 675 of their informal caregivers. Investigators will compare the effectiveness of two distinct palliative care models: a) nurse-led telephonic case management; and b) facilitated, outpatient specialty palliative care.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* English or Spanish-speaking patients ages 50 years and older
* Qualifying serious, life-limiting conditions and who are scheduled for ED discharge, observation status, or admission for two midnights or less.
* Qualifying conditions include: advanced cancer (defined as metastatic solid tumor) or poor prognosis end-stage organ failure New York Heart Association (NYHA) Class III or IV Congestive Heart Failure (CHF), End-Stage Renal Disease (ESRD), defined as Glomerular Filtration Rate (GFR) < 15 ml/min/m2 or dialysis; or Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage III or higher or stage III or IV, or oxygen-dependent chronic obstructive pulmonary disease (COPD) defined as Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Patients must have health insurance, reside within the geographical area, and have a working telephone.

Informal Caregivers:

* English or Spanish-speaking primary caregivers (relative or friend who has contact with the patient at least two times per week) ages 18 years and older.

Exclusion Criteria:

* Patients with dementia identified in the EHR, who received hospice services in the last six months, who have received 2 or more palliative care visits in the last 6 months, and those who reside in a skilled nursing or assisted living facility, or chronic care hospital.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1606 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corita R. Grudzen, MD, MSHS, FACEP, Principal Investigator — Memorial Sloan Kettering Cancer Center; Keith S. Goldfeld, DrPH, MS, MPA, Principal Investigator — NYU Langone Health
Locations (18):
- United States (18):
  - University of California, Los Angeles Ronald Reagan Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of California San Diego Medical Center, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Florida (UF), Gainesville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital/Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Health, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Troy, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health System, Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Hospital- Brooklyn, Brooklyn, New York
  - NYU Langone Health Hospital Long Island, Mineola, New York
  - Bellevue Hospital, New York, New York
  - New York University Langone Tisch Hospital, New York, New York
  - Ohio State University (OSU), Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Keith.Goldfeld@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Background] Zhao N, Cuthel AM, Storms O, Zhang R, Yamarik RL, Hill J, Kaur R, Van Allen K, Flannery M, Chang A, Chung F, Randhawa S, Alvarez IC, Young-Brinn A, Kizzie-Gillett CL, Rosini D, Isaacs ED, Hopkins E 3rd, Chan GK, Booker-Vaughns J, Maguire M, Navarro M, Pidatala NR, Dunn P, Williams P, Galvin R, Batra R, Welsh S, Vaughan W, Bouillon-Minois JB, Grudzen CR. Advancing patient-centered research practices in a pragmatic patient-level randomized clinical trial: A thematic analysis of stakeholder engagement in Emergency Medicine Palliative Care Access (EMPallA). Res Involv Engagem. 2024 Jan 23;10(1):10. doi: 10.1186/s40900-023-00539-x. PMID 38263088
- [Background] Booker-Vaughns J, Rosini D, Batra R, Chan GK, Dunn P, Galvin R, Hopkins E 3rd, Isaacs E, Kizzie-Gillett CL, Maguire M, Navarro M, Reddy Pidatala N, Vaughan W, Welsh S, Williams P, Young-Brinn A, Van Allen K, Cuthel AM, Liddicoat Yamarik R, Flannery M, Goldfeld KS, Grudzen CR. What's in This For You? What's in This For Me?: A Win-Win Perspective of Involving Study Advisory Committee Members in Palliative Care Research. J Patient Exp. 2024 Jan 2;11:23743735231224562. doi: 10.1177/23743735231224562. eCollection 2024. PMID 38188534
- [Background] Yusufov M, Adeyemi O, Flannery M, Bouillon-Minois JB, Van Allen K, Cuthel AM, Goldfeld KS, Ouchi K, Grudzen CR. Psychometric Properties of the Functional Assessment of Cancer Therapy-General for Evaluating Quality of Life in Patients With Life-Limiting Illness in the Emergency Department. J Palliat Med. 2024 Jan;27(1):63-74. doi: 10.1089/jpm.2022.0270. Epub 2023 Sep 6. PMID 37672598
- [Background] Liddicoat Yamarik R, Chiu LA, Flannery M, Van Allen K, Adeyemi O, Cuthel AM, Brody AA, Goldfeld KS, Schrag D, Grudzen CR, On Behalf Of The EMPallA Investigators. Engagement, Advance Care Planning, and Hospice Use in a Telephonic Nurse-Led Palliative Care Program for Persons Living with Advanced Cancer. Cancers (Basel). 2023 Apr 15;15(8):2310. doi: 10.3390/cancers15082310. PMID 37190238
- [Background] Brickey J, Flannery M, Cuthel A, Cho J, Grudzen CR; EMPallA Investigators. Barriers to recruitment into emergency department-initiated palliative care: a sub-study of a multi-site, randomized controlled trial. BMC Palliat Care. 2022 Feb 15;21(1):22. doi: 10.1186/s12904-021-00899-9. PMID 35168622
- [Background] Yamarik RL, Tan A, Brody AA, Curtis J, Chiu L, Bouillon-Minois JB, Grudzen CR. Nurse-Led Telephonic Palliative Care: A Case-Based Series of a Novel Model of Palliative Care Delivery. J Hosp Palliat Nurs. 2022 Apr 1;24(2):E3-E9. doi: 10.1097/NJH.0000000000000850. PMID 35149656
- [Background] Schmucker AM, Flannery M, Cho J, Goldfeld KS, Grudzen C; EMPallA Investigators. Data from emergency medicine palliative care access (EMPallA): a randomized controlled trial comparing the effectiveness of specialty outpatient versus telephonic palliative care of older adults with advanced illness presenting to the emergency department. BMC Emerg Med. 2021 Jul 12;21(1):83. doi: 10.1186/s12873-021-00478-4. PMID 34247588
- [Background] de Forcrand C, Flannery M, Cho J, Reddy Pidatala N, Batra R, Booker-Vaughns J, Chan GK, Dunn P, Galvin R, Hopkins E, Isaacs ED, Kizzie-Gillett CL, Maguire M, Navarro M, Rosini D, Vaughan W, Welsh S, Williams P, Young-Brinn A, Grudzen CR. Pragmatic Considerations in Incorporating Stakeholder Engagement Into a Palliative Care Transitions Study. Med Care. 2021 Aug 1;59(Suppl 4):S370-S378. doi: 10.1097/MLR.0000000000001583. PMID 34228019
- [Background] Tan AJ, Yamarik R, Brody AA, Chung FR, Grudzen C; EMPallA Telephonic Working Group. Development and protocol for a nurse-led telephonic palliative care program. Nurs Outlook. 2021 Jul-Aug;69(4):626-631. doi: 10.1016/j.outlook.2020.12.011. Epub 2021 Jan 21. PMID 33485590
- [Background] Grudzen CR, Schmucker AM, Shim DJ, Ibikunle A, Cho J, Chung FR, Cohen SE; EMPallA Outpatient Investigators. Development of an Outpatient Palliative Care Protocol to Monitor Fidelity in the Emergency Medicine Palliative Care Access Trial. J Palliat Med. 2019 Sep;22(S1):66-71. doi: 10.1089/jpm.2019.0115. PMID 31486726
- [Background] Grudzen CR, Shim DJ, Schmucker AM, Cho J, Goldfeld KS; EMPallA Investigators. Emergency Medicine Palliative Care Access (EMPallA): protocol for a multicentre randomised controlled trial comparing the effectiveness of specialty outpatient versus nurse-led telephonic palliative care of older adults with advanced illness. BMJ Open. 2019 Jan 25;9(1):e025692. doi: 10.1136/bmjopen-2018-025692. PMID 30813112
- [Derived] Grudzen CR, Flannery M, Van Allen K, Cuthel A, Liddicoat Yamarik R, Tan A, Cohen SE, Comstock Barker P, Brody AA, Herchek C, Siman N, Goldfeld KS; EMPallA Group. Nurse led telephonic palliative care versus specialty outpatient palliative care: pragmatic, randomised clinical trial. BMJ Med. 2025 Nov 12;4(1):e001392. doi: 10.1136/bmjmed-2025-001392. eCollection 2025. PMID 41245582
- [Derived] Maloney B, Flannery M, Bischof JJ, Van Allen K, Adeyemi O, Goldfeld KS, Cuthel AM, Chang A, Grudzen CR. Factors impacting loneliness in patients with serious life-limiting illness in the Emergency Medicine Palliative Care Access (EMPallA) study. BMC Palliat Care. 2025 Mar 8;24(1):58. doi: 10.1186/s12904-025-01699-1. PMID 40055670
- [Derived] Barker PC, Yamarik RL, Adeyemi O, Cuthel AM, Flannery M, Siman N, Goldfeld KS, Grudzen CR; EMPallA Investigators. Predictors of Specialty Outpatient Palliative Care Utilization Among Persons With Serious Illness. J Pain Symptom Manage. 2024 Dec;68(6):583-593. doi: 10.1016/j.jpainsymman.2024.08.004. Epub 2024 Aug 22. PMID 39179000

RESULTS

PARTICIPANT FLOW:
Groups:
- Nurse-led Telephonic Case Management (Patients Only): * Telephonic nurses will contact patients within 72 hours of enrollment
  * Patients will speak with the telephonic nurse over the phone once a week (or as often as needed) for a duration of 6 months.
  Nurse-led telephonic case management: Telephonic meetings with a palliative care nurse. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
- Nurse-led Telephonic Case Management (Caregivers Only): Caregivers of patients enrolled in the nurse-led telephonic case management arm.
- Facilitated, Outpatient Specialty Palliative Care (Patients Only): * Patients will be scheduled for their first in-person palliative care visit within two weeks of enrollment and then once a month for 6 months.
  * Clinic visits will be scheduled the same day as other specialty appointments if possible
  Facilitated,outpatient specialty palliative care: In-person or telehealth palliative care visits with a palliative care provider. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
- Facilitated, Outpatient Specialty Palliative Care (Caregivers Only): Caregivers of patients in the facilitated, outpatient specialty palliative care arm.
Period: Overall Study
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Started | 639 | 155 | 644 | 168
Completed | 418 | 93 | 409 | 108
Not Completed | 221 | 62 | 235 | 60
Not completed — Lost to Follow-up | 122 | 26 | 141 | 28
Not completed — Death | 99 | 36 | 94 | 32

BASELINE CHARACTERISTICS:
Groups:
- Nurse-led Telephonic Case Management (Caregiver Only): Caregivers of patients enrolled in the nurse-led telephonic case management arm.
- Facilitated, Outpatient Specialty Palliative Care (Caregivers Only): Caregivers of patients enrolled in the facilitated, outpatient specialty palliative care arm.
- Total: Total of all reporting groups
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Nurse-led Telephonic Case Management (Caregiver Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only) | Total
Number analyzed (Participants) | 541 | 119 | 549 | 136 | 1345
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10) | 55.8 (15.7) | 66.6 (10.2) | 56.8 (13.7) | 61.4 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 303 | 81 | 284 | 89 | 757
  Male | 238 | 36 | 265 | 47 | 586
  Unknown/Missing | 0 | 2 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 9 | 73 | 20 | 152
  Not Hispanic or Latino | 482 | 108 | 469 | 115 | 1174
  Unknown or Not Reported | 9 | 2 | 7 | 1 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 4 | 0 | 10
  Asian | 7 | 2 | 3 | 1 | 13
  Native Hawaiian or Pacific Islander | 3 | 1 | 4 | 0 | 8
  Black or African American | 189 | 34 | 170 | 33 | 426
  White | 288 | 71 | 307 | 86 | 752
  More than one race | 7 | 0 | 11 | 0 | 18
  Other race | 38 | 8 | 41 | 14 | 101
  Missing | 5 | 1 | 9 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 541 | 119 | 549 | 136 | 1345

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life for Patients, as Measured by the Functional Assessment of Cancer Therapy - General (FACT-G)
Description: * Measured by change from enrollment to 6 months
  * Used to measure a person's quality of life
  * 27 questions total
  * 5-point Likert scale
  * Reverse code select items per scoring guidelines at facit.org, then calculate a summary score for each respondent. The total score ranges from 0-108 points; higher scores indicate greater quality of life.
Time Frame: Baseline, Month 6
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 416 | 408
score on a scale | 3.7 (14.6) | 3.1 (15)

2. Secondary Outcome: Number of Emergency Department (ED) Revisits
Description: Measured from enrollment to 12 months as a count of ED revisits, via self-report and EHR abstraction.
Time Frame: Up to Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Revisits
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 639 | 644
Revisits | 2.5 (3.5) | 2.7 (3.8)

3. Secondary Outcome: Number of Inpatient Days
Description: Measured from enrollment to 12 months as the number of inpatient days, via self-report and EHR extraction.
Time Frame: Up to Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 639 | 644
Days | 8.1 (15.3) | 8.6 (18.6)

4. Secondary Outcome: Proportion of Participants Who Used Hospice
Description: Measured from enrollment to 12 months as the proportion of participants who used hospice, via self-report and EHR abstraction.
Time Frame: Up to Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Number; unit: Proportion of participants
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 635 | 641
Proportion of participants | 0.16 | 0.18

5. Secondary Outcome: Change in Loneliness, as Measured by the Three-Item Loneliness Scale
Description: * Used to measure how often a person feels disconnected from others
  * Three questions total
  * 3-point rating scale (1 = Hardly ever, 2 = Some of the time, 3 = Often)
  * Total score is the sum of responses and ranges from 3 to 9; higher scores indicate greater loneliness.
  * measured by change from enrollment to 3 months
Time Frame: Baseline, Month 3
Population: Caregivers were not assessed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 466 | 442
score on a scale | 0 [-1 to 1] | 0 [-1 to 1]

6. Secondary Outcome: Change in Loneliness, as Measured by the Three-Item Loneliness Scale
Description: * Used to measure how often a person feels disconnected from others
  * Three questions total
  * 3-point rating scale (1 = Hardly ever, 2 = Some of the time, 3 = Often)
  * Total score is the sum of responses and ranges from 3 to 9; higher scores indicate greater loneliness.
  * measured by change from enrollment to 6 months
Time Frame: Baseline, Month 6
Population: Caregivers were not assessed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 410 | 405
score on a scale | 0 [-1 to 1] | 0 [-1 to 1]

7. Secondary Outcome: Change in Loneliness, as Measured by the Three-Item Loneliness Scale
Description: * Used to measure how often a person feels disconnected from others
  * Three questions total
  * 3-point rating scale (1 = Hardly ever, 2 = Some of the time, 3 = Often)
  * Total score is the sum of responses and ranges from 3 to 9; higher scores indicate greater loneliness.
  * measured by change from enrollment to 12 months
Time Frame: Baseline, Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 334 | 321
score on a scale | 0 [-1 to 1] | 0 [-1 to 1]

8. Secondary Outcome: Change in Symptom Burden, as Measured by Edmonton Symptom Assessment Scale Revised (ESAS-r)
Description: * Used to measure severity of symptoms
  * 10 questions
  * Each item is rated on a 0-10 scale (0= none to 10 worst possible)
  * Total score ranges from 0 to 100; higher scores indicate greater severity of symptoms.
  * measured by change from enrollment to 3 months
Time Frame: Baseline, Month 3
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 471 | 447
score on a scale | -3.8 (12.1) | -3.3 (12.2)

9. Secondary Outcome: Change in Symptom Burden, as Measured by Edmonton Symptom Assessment Scale Revised (ESAS-r)
Description: * Used to measure severity of symptoms
  * 10 questions
  * Each item is rated on a 0-10 scale (0= none to 10 worst possible)
  * Total score ranges from 0 to 100; higher scores indicate greater severity of symptoms.
  * measured by change from enrollment to 6 months
Time Frame: Baseline, Month 6
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 413 | 407
score on a scale | -3 (12.7) | -2.5 (12.9)

10. Secondary Outcome: Change in Symptom Burden, as Measured by Edmonton Symptom Assessment Scale Revised (ESAS-r)
Description: * Used to measure severity of symptoms
  * 10 questions
  * Each item is rated on a 0-10 scale (0= none to 10 worst possible)
  * Total score ranges from 0 to 100; higher scores indicate greater severity of symptoms.
  * measured by change from enrollment to 12 months
Time Frame: Baseline, Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 339 | 323
score on a scale | -3.3 (13) | -1.9 (13.4)

11. Secondary Outcome: Change in Caregiver Physical Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: * Quality of life for informal caregivers will be measured using the 10-item Patient-Reported Outcome Measurement Information System (PROMIS-10), an instrument designed to measure perceptions of health using global health items. It contains a global physical health scale and a global mental health scale.
  * Scored by reverse coding with a raw score ranging from 0-20; 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health. Scales are scored using the raw sum to T-score tables for physical health and mental health. T-scores range from 0-100; higher scores reflect better functioning.
  * measured by change from enrollment to 3 months
Time Frame: Baseline, Month 3
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Nurse-led Telephonic Case Management (Caregivers Only): * Telephonic nurses will contact patients within 72 hours of enrollment
  * Patients will speak with the telephonic nurse over the phone once a week (or as often as needed) for a duration of 6 months.
  Nurse-led telephonic case management: Telephonic meetings with a palliative care nurse. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
- Facilitated, Outpatient Specialty Palliative Care (Caregivers Only): * Patients will be scheduled for their first in-person palliative care visit within two weeks of enrollment and then once a month for 6 months.
  * Clinic visits will be scheduled the same day as other specialty appointments if possible
  Facilitated,outpatient specialty palliative care: In-person or telehealth palliative care visits with a palliative care provider. Palliative care is specialized medical care focused on providing a personalized layer of support dedicated to helping patients and their families cope with a serious illness.
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 106 | 119
score on a scale | -0.3 (5.2) | -0.6 (4.4)

12. Secondary Outcome: Change in Caregiver Physical Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: * Quality of life for informal caregivers will be measured using the 10-item Patient-Reported Outcome Measurement Information System (PROMIS-10), an instrument designed to measure perceptions of health using global health items. It contains a global physical health scale and a global mental health scale.
  * Scored by reverse coding with a raw score ranging from 0-20; 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health. Scales are scored using the raw sum to T-score tables for physical health and mental health. T-scores range from 0-100; higher scores reflect better functioning.
    * measured by change from enrollment to 6 months
Time Frame: Baseline, Month 6
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 93 | 107
score on a scale | 0.1 (5.2) | -0.3 (4.4)

13. Secondary Outcome: Change in Caregiver Physical Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: * Quality of life for informal caregivers will be measured using the 10-item Patient-Reported Outcome Measurement Information System (PROMIS-10), an instrument designed to measure perceptions of health using global health items. It contains a global physical health scale and a global mental health scale.
  * Scored by reverse coding with a raw score ranging from 0-20; 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health. Scales are scored using the raw sum to T-score tables for physical health and mental health. T-scores range from 0-100; higher scores reflect better functioning.
    * measured by change from enrollment to 12 months
Time Frame: Baseline, Month 12
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 77 | 77
score on a scale | -0.8 (5.6) | -0.2 (5.1)

14. Secondary Outcome: Caregiver Bereavement, as Measured by the Texas Inventory of Grief
Description: * Measured at 3 months post-patient death
  * Used to measure a caregiver's bereavement
  * 19 items; each rated on a 5-point scale from 0 (never) to 4 (always)
  * Total score is the sum of responses and ranges from 0 to 76; higher scores indicate greater levels of grief
Time Frame: 3 Months Post-Patient Death
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 34 | 29
score on a scale | 31.2 (9.8) | 29.3 (8.7)

15. Secondary Outcome: Change in Caregiver Strain, as Measured by the Zarit Burden Interview (ZBI-12)
Description: * Measured as change from enrollment to Month 3
  * Used to measure a caregiver's strain
  * 12 items; each rated on a 3-point scale from 0 (yes, on a regular basis) to 3 (no)
  * Total score is the sum of responses and ranges from 0 to 48; higher scores indicate greater burden
Time Frame: Baseline, Month 3
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 108 | 120
score on a scale | -0.5 (6.9) | -0.6 (6.3)

16. Secondary Outcome: Change in Caregiver Strain, as Measured by the Zarit Burden Interview (ZBI-12)
Description: * Measured as change from enrollment to Month 6
  * Used to measure a caregiver's strain
  * 12 items; each rated on a 3-point scale from 0 (yes, on a regular basis) to 3 (no)
  * Total score is the sum of responses and ranges from 0 to 48; higher scores indicate greater burden
Time Frame: Baseline, Month 6
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 93 | 108
score on a scale | -0.6 (7.3) | 1.3 (5.9)

17. Secondary Outcome: Change in Caregiver Strain, as Measured by the Zarit Burden Interview (ZBI-12)
Description: * Measured as change from enrollment to Month 12
  * Used to measure a caregiver's strain
  * 12 items; each rated on a 3-point scale from 0 (yes, on a regular basis) to 3 (no)
  * Total score is the sum of responses and ranges from 0 to 48; higher scores indicate greater burden
Time Frame: Baseline, Month 12
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 75 | 78
score on a scale | -0.9 (6.5) | 1 (7.7)

18. Secondary Outcome: Change in Quality of Life for Patients, as Measured by the FACT-G
Description: * Measured by change from enrollment to 3 months
  * Used to measure a person's quality of life
  * 27 questions total
  * 5-point Likert scale
  * Reverse code select items per scoring guidelines at facit.org, then calculate a summary score for each respondent. The total score ranges from 0-108 points; higher scores indicate greater quality of life.
Time Frame: Baseline, Month 3
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 470 | 452
score on a scale | 3.4 (14.2) | 3.6 (14.6)

19. Secondary Outcome: Change in Quality of Life for Patients, as Measured by the FACT-G
Description: * Measured by change from enrollment to 12 months
  * Used to measure a person's quality of life
  * 27 questions total
  * 5-point Likert scale
  * Reverse code select items per scoring guidelines at facit.org, then calculate a summary score for each respondent. The total score ranges from 0-108 points; higher scores indicate greater quality of life.
Time Frame: Baseline, Month 12
Population: Caregivers were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only)
Number analyzed (Participants) | 337 | 328
score on a scale | 4 (17.2) | 3.7 (15.5)

20. Secondary Outcome: Change in Caregiver Mental Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: as for outcome 11
Time Frame: Baseline, Month 3
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 106 | 118
score on a scale | 0.2 (7.9) | 0.3 (7.9)

21. Secondary Outcome: Change in Caregiver Physical Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: as for outcome 12
Time Frame: Baseline, Month 6
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 93 | 106
score on a scale | 1.6 (7.4) | -0.1 (6.6)

22. Secondary Outcome: Change in Caregiver Physical Health Quality of Life, as Measured by the Patient-Reported Outcome Measurement Information System (PROMIS-10)
Description: as for outcome 12
Time Frame: Baseline, Month 12
Population: Patient participants were not assessed for this outcome measure; only Caregiver participants were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
Number analyzed (Participants) | 75 | 76
score on a scale | -0.5 (6.9) | 0.8 (7.9)

ADVERSE EVENTS:
Time Frame: 12 months
Description: An Adverse Event (AE) would be reportable if discussion surrounding end-of-life issues or processes causes a patient or caregiver severe emotional distress as confirmed by the site PI. PM to monitor and inform mPIs of any AEs or harmful, unexpected Severe AEs related to the research. The mPIs and Co-Is were versed in these reporting procedures (required for all research conducted at each respective site).
Groups:
- Nurse-led Telephonic Case Management (Caregivers Only): Caregivers of patients in the nurse-led telephonic case management arm.
Arm/Group | Nurse-led Telephonic Case Management (Patients Only) | Nurse-led Telephonic Case Management (Caregivers Only) | Facilitated, Outpatient Specialty Palliative Care (Patients Only) | Facilitated, Outpatient Specialty Palliative Care (Caregivers Only)
All-Cause Mortality (participants affected / at risk) | 99/639 | 36/155 | 94/644 | 32/168
Serious Adverse Events (participants affected / at risk) | 0/639 | 0/155 | 0/644 | 0/168
Other Adverse Events (participants affected / at risk) | 0/639 | 0/155 | 0/644 | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03325985/Prot_SAP_000.pdf